CLINICAL TRIAL: NCT06892184
Title: Importance of the Type of Communication Used During Paraapical Anesthesia in Dentistry: Randomized Clinical Trial
Brief Title: Importance of the Type of Communication Used During Paraapical Anesthesia in Dentistry
Acronym: CADA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RBHP 2024 MELIN (CADA); 2024-A02606-41 (Other: 2024-A02606-41)
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Communication Skills; Dental Care; Hypnosis
Keywords: Therapeutic communication; Dental care; Induced pain; Nocebo effect; hypnosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hypnotic communication (Experimental)
  Interventions: Behavioral: hypnotic communication
- conventional communication (Active Comparator)
  Interventions: Behavioral: conventional communication

INTERVENTIONS:
Behavioral: hypnotic communication — During local anaesthesia, the operator will not remain silent, nor will he describe to his patient the anaesthesia he is performing, nor warn his patient of possible future pain. When performing anesthesia, the operator will use a dissociative, hypnotic language, standardized across all patients.
  Arms: hypnotic communication
Behavioral: conventional communication — suggestions typically uttered by the practitioner, who describes what he is doing and warns of possible pain.
  Arms: conventional communication

SUMMARY:
Can we improve our communication to provide better care for our patients? In the healthcare field, the patient's experience is closely linked to pain management. The dental profession often requires simple but invasive procedures, such as local anaesthetics for example, which are providers of discomfort and anxietý that cannot be ignored. Fear of the dentist or dental care is a widespread phenomenon in the general population, since dental anxiety is estimated to affect 36% of the population, and 12% are thought to suffer from extreme fear. Clinicians traditionally warn patients of pain before para-apical anesthesia. This is not surprising, since even today, during initial training for practitioners, patients are taught to be informed, or even warned, of the pain to come, for ethical reasons (i.e., not to lie to the patient) and "so that he/she can prepare for it" (what we will refer to in the remainder of this protocol as classic communication). In the same way as when the patient has acute or induced pain, as is the case here (pain induced by the anesthetic injection), the practitioner also learns to ask if the patient is in pain, and how much. However, the use of pain-related words or a focus on pain can lead to significant anxiety, which in turn lowers the pain threshold. Conversely, the use of positive communication is important, as it can improve the patient's perception of pain and subjective experience. There is a body of literature on the impact of hypnotic communication on pain during painful treatment, but in fields other than dentistry (e.g. venous voice placement - Fusco 2020). To our knowledge, there is no scientific basis on the impact of the type of communication on patient pain in the field of dentistry. If, as we assume, we do indeed find similar results in other fields of medicine, this basis could serve as a basis for modifying the teaching and hence the practice of our young practitioners. We aim to compare the effects of two types of communication (hypnotic and conventional) on patients' pain, comfort and anxiety during para-apical anesthesia in dentistry. Anxiety and comfort were assessed prior to anesthesia on a numerical scale ranging from 0 (no anxiety or comfort) to 10 (greatest imaginable anxiety or comfort). This assessment of anxiety and comfort is asked again after anesthesia has been performed, as well as the pain experienced during anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient over 18 years of age requiring para-apical anesthesia for dental care.
* Patient informed of the constraints of the study and having given written consent.
* Patient covered by social security.
* Patient with a good command of French.

Exclusion Criteria:

* Pregnant or breastfeeding women, or women who may become pregnant.
* Patients under 18 years of age.
* Patients presenting to the department in an emergency situation (which may increase stress).
* Any medical condition deemed by the investigator to be incompatible with the study.
* Known hypersensitivity to amide-bonded local anesthetics or to any of the excipients.
* Anticoagulant treatment or known blood crase disorders.
* Porphyrias.
* Atrioventricular conduction disorders requiring permanent electrosystolic training not yet performed.
* Epilepsy not controlled by treatment.
* Patient uncooperative, unable to speak or read French fluently, unable to understand the principle of a pain scale, unable to understand the study or unable to sign informed consent.
* Patients under guardianship, curatorship or deprived of liberty.
* Patients premedicated with anxiolytics
* Care requiring anesthesia other than para-apical anesthesia
* Patient highly anxious about dental treatment (Score ≥15 on Corah scale)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
pain intensity | assessed just after anesthesia
  Perception of pain experienced by the patient during anesthesia, assessed after anesthesia by numerical scale from 0 to 10.

SECONDARY OUTCOMES:
Self-assessment of comfort | before and after anesthesia
  numerical scale from 0 to 10
Self-assessment of anxiety | before and after anesthesia
  numerical scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Céline Melin, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No